CLINICAL TRIAL: NCT01428362
Title: A Randomized, Placebo-Controlled, Double-Blind, Crossover Study to Evaluate the Safety, Tolerability and Efficacy of VI-1121 in Subjects With Alzheimer's Disease
Brief Title: VI-1121 for the Treatment Alzheimer's Disease
Acronym: AD-201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AD-201
Record Dates: First submitted 2011-08-31; First posted 2011-09-05 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-11

CONDITIONS: Alzheimer's Disease
Keywords: donepezil; VI-1121
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo/VI-1121 (Experimental): Subjects received placebo during first treatment period and active treatment with VI-1121 during the second treatment period.
  Interventions: Drug: VI-1121; Drug: Placebo
- VI-1121/Placebo (Experimental): Subjects received active treatment with VI-1121 during the first treatment period and placebo during the second treatment period.
  Interventions: Drug: VI-1121; Drug: Placebo

INTERVENTIONS:
Drug: VI-1121
Drug: Placebo

SUMMARY:
The purpose of this study is to determine whether VI-1121 is safe, well tolerated, and effective as a daily treatment for Alzheimer's disease that is worsening despite current treatment.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Alzheimer's disease
* CT or MRI within 2 years prior to study
* stable dose of current Alzheimer's treatment for at least 3 months

Exclusion Criteria:

* advanced, severe, progressive or unstable disease
* history of cerebrovascular disease or myocardial infarction within 6 months

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is the change in Alzheimer's Disease Assessment-Cognitive Subscale (ADAS-Cog) score from baseline to Week 12 of each treatment period. | 12 weeks

SECONDARY OUTCOMES:
The secondary efficacy endpoint is the mean change in Mini-Mental State Examination (MMSE) score from baseline to Week 12 of each treatment period. | 12 weeks
Percentage of subjects who achieve 3-point improvement in ADAS-Cog score from baseline to Week 12 of each treatment period. | 12 Weeks
Change in Clinician's Interview Based Impression of Change Plus Caregiver's Input (CIBIC-plus) score from baseline to Week 12 of each treatment period | 12 Weeks
Mean change in Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) score from baseline to Weeks 4, 8, and 12 of each treatment period | 4, 8, and 12 Weeks

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - San Francisco, California
  - Santa Monica, California
  - Sunrise, Florida
  - Louisville, Kentucky
  - Las Vegas, Nevada
  - Toms River, New Jersey
  - New Windsor, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Toledo, Ohio
  - Plano, Texas